CLINICAL TRIAL: NCT05746663
Title: Kronik Ayak Bileği İnstabilitesi Olan Voleybolcularda Denge ve Patlayıcı Güç Üzerine Morfolojik Bir Çalışma
Brief Title: A Morphological Study in Volleyball Athletes With Cronic Ankle Instability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: GO 22/885
Record Dates: First submitted 2023-01-30; First posted 2023-02-28 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Ankle Injuries; Instability; Ankle (Ligaments) (Old Injury); Radiological Devices Associated With Adverse Incidents, Diagnostic and Monitoring Devices; Athlete Foot
MeSH Terms: conditions — Ankle Injuries; Disease; Tinea Pedis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The former purpose of this study to investigate the effect of transverse abdominis, lumbar multifidus, vastus lateralis, lateral gastrocnemius, anterior talofibular ligament of morphology on explosive power and balance performance in cronic ankle instability with volleyball players. The latter purpose of this study to determine morphological characteristics volleyball players with and without cronic ankle insatbility of trunk muscle morphology, field tests and the muscle morphology features between the body affected and unaffected sides whose those with chronic ankle instability.This study was designed as a cross-sectional. Twelve volleyball players with chronic ankle instability who meet the criteria determined by the ankle consortium will be included in study group. Twelve asymptomatic volleyball players who have been training at least three days a week for at least one year will be include in the control group. They will consist of 24 volleyball players between 14-35 years of age.Morphological characteristics of anterior talofibular ligament, transverse abdominis, lumbar multifidus, vastus lateralis, lateral gastrocnemius will be evaluated via ultrasound, explosive power with squat jump, counter movement jump and balance performance by Y-Balance Test. Trunk muscle morphology, core stabilization, explosive power, balance performance will have been compered in volleyball players with and without chronic ankle instability. The effects of morphological features on explosive power and balance performance will have been determined. It is anticipated that by determining the parameters that can be affected by instability with volleyball players, it will guide the professionals working in the field, countribute to treatment and preventive treatment programs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion for the CAI group followed the International Ankle Consortium guidelines.

Criteria for inclusion in the control group:

To train for 1 hour at least 3 days a week for at least 1 year, Cumberland Ankle Instability Instrument (CAIT) score of 25 or higher, To have a Tegner activity level of 4 and above, It is not to have a systemic disease

Exclusion Criteria:

The patient will be excluded from the study in the event of the presence of at least one of the following criteria:

Having undergone ankle, knee, hip surgery, Having bilateral ankle instability, Having suffered a known musculoskeletal injury of the hip Having suffered an ankle sprain during the evaluation process

Criteria for exclusion from the study:

Withdraw to any period

Ages: 14 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Hacettepe University will be directed from the referred athletes.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-09-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Muscle morphology | 1 day
  Morphological characteristics of anterior talofibular ligament, transverse abdominis, lumbar multifidus, vastus lateralis, lateral gastrocnemius will be evaluated via ultrasound imaging
Balance | 1 day
  Y Balance Test
Expolsive Power | 1 day
  Squat jump, Countermovement jump Test
Core stability | 1 day
  Sharmannn's Core Stability Tet

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Aynur Demirel, Ankara, Turkey (Türkiye)